CLINICAL TRIAL: NCT02787993
Title: Feasibility and Acceptability of a Behavioral Symptom Management Program for Patients With Advanced Breast Cancer in Singapore and the US
Brief Title: ICAN Symptoms Duke-NUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00072023
Record Dates: First submitted 2016-05-24; First posted 2016-06-02 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Mutli-Symptom management(CBT) (Active Comparator): Learn to manage distress, fatigue, and/or pain via (Cognitive Behavioral Multi-Symptom management (CBT) four one hour sessions.
  Interventions: Behavioral: Cognitive Behavioral Mult-Symptom management(CBT)
- Treatment as usual (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Cognitive Behavioral Mult-Symptom management(CBT) — Learn to manage distress, fatigue, and/or pain via Cognitive Behavioral Multi-Symptom Management(CBT). Four sessions will be conducted each session is approximately one hour.
  Arms: Cognitive Behavioral Mutli-Symptom management(CBT)

SUMMARY:
The purpose of this study is to conduct a pilot randomized controlled trial (RCT) to examine the feasibility, acceptability, and cultural sensitivity of a cross-cultural cognitive behavioral therapy (CBT) multi-symptom management protocol targeting distress (anxiety, depression), pain, and fatigue in women with advanced stage breast cancer in Singapore and the US.

DETAILED DESCRIPTION:
Up to two-thirds of women with advanced breast cancer experience significant symptom burden (e.g., distress, pain, fatigue), yet these symptoms are not adequately addressed. Cognitive behavioral therapy (CBT) protocols designed to teach patients strategies to improve their symptom management may be helpful in alleviating multiple symptoms. The efficacy of CBT protocols for reducing distinct symptoms in early-stage breast cancer has been shown in Western countries; however, the role of CBT protocols for multiple symptoms in late-stage cancer is less clear. This study aims to investigate the feasibility and acceptability and obtain estimates of efficacy of a novel, cross-cultural multi-symptom (i.e., anxiety and depression, pain, fatigue) CBT protocol in advanced breast cancer patients. A randomized controlled design will compare patients receiving the CBT protocol to a waitlist control condition in both Singapore and United States patients. The goal of this collaborative effort is to determine the scalability of the cross- cultural intervention. This IRB protocol only represents the Duke US portion of the project; Duke-NUS will obtain their own IRB approvals.

ELIGIBILITY:
Inclusion Criteria:

* being at least 21 years of age
* a diagnosis of stage IV breast cancer
* being able and willing to attend study appointments
* being able to speak/read English
* estimated survival of at least 3 months.

Exclusion Criteria:

* they have an active serious mental illness (e.g., schizophrenia, bipolar disorder) as indicated by medical records
* if visual, hearing, or cognitive impairment will interfere with intervention.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by study accrual by meeting recruitment goal | 6 weeks
  Feasibility will be shown by meeting targeted study accrual (N=40) in the 12-month study period.
Feasibility as measured by study attrition which will be assessed by patients who do not complete the post-assessment. | 6 weeks
  Feasibility will be shown by no more than 20% study attrition.
Feasibility as measured by adherence to the study protocol by number of intervention sessions completed by the participant | 6 weeks
  Feasibility will be shown by adherence to at least 75% of the intervention sessions (3/4)
Acceptability, as measured by Client Satisfaction Questionnaire 10-item version | 6 weeks
  Acceptability will be indicated by at least 80% of the participants reporting satisfaction with the CBT protocol (mean score of 7) on the CSQ
Cultural Sensitivity | 6 weeks
  Quantitative data will be collected with a 5-minute verbal interview to the participant inquiring about cultural relevance and sensitivity.

SECONDARY OUTCOMES:
Change in anxiety and depression | Baseline and 6 weeks
  The Hospital Anxiety and Depression Scale14 will be used to assess distress (anxiety and depressive symptoms)
Change in pain | Baseline and 6 weeks
  Pain will be assessed with the Brief Pain Inventory (BPI)
Change in fatigue | Baseline and 6 weeks
  Fatigue will be assessed with the PROMIS Adult Fatigue Profile Short Form.
Change in Pain | Baseline and 6 weeks
  Pain will be assessed with the Pain Disability Index

CONTACTS AND LOCATIONS:
Overall Officials: Tamara J Somers, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States